CLINICAL TRIAL: NCT04569318
Title: A Study To Assess A Novel Form Of Cataract Treatment Using The Non-Invasive REVISYON Proof-Of-Concept Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edinburgh Biosciences Ltd (Industry)
Collaborators: Onorach Clinical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EB-14-LAT
Record Dates: First submitted 2020-09-17; First posted 2020-09-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Single arm interventional study
Masking Description: Unmasked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Treatment with treatment beam.
  Interventions: Device: Treatment Beam

INTERVENTIONS:
Device: Treatment Beam — One of the subject's eyes will be treated with the treatment beam (20mW) up to 8 times for 15 minutes.

SUMMARY:
Single arm proof-of-concept trial to evaluate the safety and efficacy of the REVISYON PoC Device in the treatment of cataract.

DETAILED DESCRIPTION:
Single arm, single site proof-of-concept trial to evaluate the safety and efficacy of the REVISYON PoC Device, with 8 x 15-minute twice-weekly treatments and 3 month safety follow-up, in the treatment of cataract.

Only one of the subject's eyes will be treated during the study. In addition, spectral data (fluorescent emission) will be collected using the device to monitor the progress of the treatment, and to determine the suitability of these measurements for future clinical diagnoses

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with nuclear sclerotic (NS) lens opacities cataract, LOCS III grade 1 to 3 (moderate), as confirmed by the Investigator
2. Subject aged between 55 and 85 years of age (inclusive) at the time of consent
3. Best corrected visual acuity (BCVA) of 0.3 or worse due to cataract only
4. Subject whom the medical health history has been reviewed by the Investigator and medical records do not contraindicate the participation to the study
5. Subject who is judged suitable for the study after ophthalmic examination carried out by the Investigator
6. Be able and willing to follow instructions, including participation in all study assessments and visits, according to the opinion of the investigator - including being able to sit upright for at least 20 mins (duration of the treatment)

Exclusion Criteria:

1. Subject unable to give voluntary written informed consent, is unlikely to cooperate or is legally incompetent, including subjects who are institutionalised by court or official order, or in a dependency relationship with sponsor, testing centre or investigator
2. Subject who had been clinically diagnosed with any eye diseases which may impact upon the treatment, or the subject's ability to be assessed after treatment
3. Subject with shallow anterior chamber
4. Subject who have had a fluorescence angiogram or any use of fluorescein within the last 3 days
5. Subject presenting eye infection or eye damage in either eye
6. Subject routinely using contact lenses
7. Planned replacement of crystalline lens with intraocular lens (IOL) implant within the planned study period
8. Any condition which could interfere with the subject's ability to comply with the study including participation in all study assessments and visits.
9. Subject who had undergone a treatment using photodynamic drugs within the last 30 days. (Including but not limited to methylene blue, toluidine blue, Visudyne®, Foscan, Photofrin or 5-aminolevulinic acid/ALA)
10. Subject diagnosed with any other health condition which, in the opinion of the Investigator, would pose a safety risk to the subject by participating in the study, or may interfere with or jeopardise the study evaluation, procedures or completion
11. Subject currently receiving treatment in another investigational study or has completed another investigational study within the last 30 days
12. Females who are pregnant or lactating
13. Females who are of childbearing potential (menses within the last 12 months) and not taking adequate contraceptive precautions are excluded from the trial. Females of childbearing potential taking acceptable contraceptive precautions may be included.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Safety: assessed by changes in the Local Ocular Tolerability (LOT) Visual Analogue Scale (VAS) | 20 weeks
  Assessment of safety defined as changes in the LOT VAS. A self-administered 7-item (foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision, photophobia) 100 mm VAS on which 0 means no symptoms and 100 means the worst possible discomfort. VAS Ocular Tolerability Overall score is the mean of all VAS Ocular Tolerability symptom scores per visit per eye
Efficacy: Cataract Grade | 5 weeks
  Assessment of efficacy, defined as treating cataract assessed using Lens Opacities Classification System (LOCS) III. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in cataract severity | 5 weeks
  Assessed using Objective Scatter Index (OSI) using Visiometrics HD Analyser. Higher scores mean a worse outcome.
Change in visual acuity | 5 weeks
  Assessed using LogMAR (Logarithm of the Minimum Angle of Resolution) scale. Higher scores mean a worse outcome.
Change in light scatter | 5 weeks
  Assessed using Visiometrics HD Analyser. Higher scores mean a worse outcome.
Change in functional impairment due to cataract | 5 weeks
  Assessed using VF-14 (Visual Function Index) questionnaire data. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Executive, Study Chair — Edinburgh Biosciences Ltd
Locations (1):
- Dr.Solomatina Acu Centrs, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No